CLINICAL TRIAL: NCT04295772
Title: A Phase 2 Clinical Study to Evaluate the Pharmacokinetics, Safety, and Efficacy of Doravirine/Islatravir in Pediatric Participants With HIV-1 Infection Who Are Virologically Suppressed or Treatment-Naïve, Are Less Than 18 Years of Age, and Weigh Greater Than or Equal to 35 kg
Brief Title: Doravirine/Islatravir (DOR/ISL) in Pediatric Participants With Human Immunodeficiency Virus Type 1 (HIV-1) Who Are <18 Years of Age and Weigh ≥35 kg (MK-8591A-028)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8591A-028; MK-8591A-028 (Other: Merck Protocol Number); 2019-003597-10 (EudraCT Number)
Record Dates: First submitted 2020-03-03; First posted 2020-03-04 (Actual); Results first posted 2023-02-24 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — doravirine; islatravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DOR/ISL (Experimental): Pediatric participants with HIV-1 infection receive DOR/ISL for 96 weeks.
  Interventions: Drug: DOR/ISL

INTERVENTIONS:
Drug: DOR/ISL — 100 mg DOR/0.75 mg ISL FDC tablet taken once daily by mouth.
  Other Names: MK-8591A; Doravirine/islatravir

SUMMARY:
This is a phase 2, single-group, multi-site, open-label study of an islatravir/doravirine (ISL/DOR, MK-8591A) fixed dose combination (FDC) for the treatment of human immunodeficiency virus type 1 (HIV-1) infection in pediatric participants who are virologically suppressed (VS) on antiretroviral therapy (ART) for ≥3 months or are treatment-naive (TN). The primary purposes of the study are 1) to examine the steady-state pharmacokinetics (PK) of ISL in plasma; 2) the steady-state PK of ISL-triphosphate (ISL-TP) in peripheral blood mononuclear cells (PBMCs); and 3) to examine the safety and tolerability of ISL/DOR.

DETAILED DESCRIPTION:
As of protocol amendment 03 (approved 08-Feb-2022), all participants have been discontinued from study therapy and will be switched to non-study antiretroviral therapy and monitored for safety. The present results cover data obtained through the cut-off date of 30-Mar-2022, and will be updated once monitoring is completed.

ELIGIBILITY:
Inclusion Criteria:

* Is HIV-1 positive, is <18 years of age, and weighs ≥35 kg at screening.
* VS Participants: Is HIV-1 positive at Screening with plasma HIV-1 RNA <50 copies/mL and has been receiving continuous, stable oral 2-drug or 3-drug combination ART ± PK booster with documented viral suppression for ≥3 months prior to providing documented informed consent/assent and has no history of prior virologic treatment failure on any past or current regimen.
* TN Participants: Is HIV-1 positive at Screening with plasma HIV-1 RNA ≥500 copies/mL and is naive to ART defined as having received <=10 days of prior therapy with any antiretrovirals following HIV-1 diagnosis other than pre-exposure prophylaxis (PrEP) or potentially exposed person (PEP).
* If female, is not pregnant or breastfeeding, and is either 1) not a woman of childbearing potential (WOCBP) or 2) is a WOCBP and is using acceptable contraception or is abstinent.

Exclusion Criteria:

* Has HIV-2 infection.
* Has hypersensitivity or other contraindication to any of the components of the study drugs as determined by the investigator.
* Has an active diagnosis of hepatitis due to any cause, including active hepatitis B virus (HBV) infection (defined as hepatitis B surface antigen [HBsAg]-positive or HBV deoxyribonucleic acid [DNA] positive).
* Has a history of malignancy ≤5 years prior to providing documented informed consent except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or cutaneous Kaposi's sarcoma.
* Has a history or current evidence of any condition (including active tuberculosis infection), therapy, laboratory abnormality or other circumstance (including drug or alcohol use or dependence) that might, in the opinion of the investigator, confound the results of the study or interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate.
* Is taking or is anticipated to require systemic immunosuppressive therapy, immune modulators, or any prohibited therapies from 45 days prior to Day 1 through the study treatment period.
* Is currently taking long-acting cabotegravir-rilpivirine.
* Is currently participating in or has participated in an interventional clinical study with an investigational compound or device from 45 days prior to Day 1 through the study treatment period.
* Has a documented or known virologic resistance to DOR/ISL (DOR resistance substitutions in reverse transcriptase: V106A/M, V108I, Y188L, H221Y, P225H, F227C/L, M230I/L, L234I, P236L, or Y318F; ISL resistance substitution in reverse transcriptase: M184V/I).
* Has exclusionary laboratory values.
* Is female and expecting to conceive or donate eggs at any time during the study.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2023-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (17):
- United States (4):
  - Children's National Medical Center ( Site 1816), Washington D.C., District of Columbia
  - Emory Children's Center ( Site 1805), Atlanta, Georgia
  - Johns Hopkins University ( Site 1800), Baltimore, Maryland
  - Duke University ( Site 1807), Durham, North Carolina
- Italy (2):
  - Azienda Ospedaliera Luigi Sacco ( Site 1300), Milan
  - IRCCS Ospedale Pediatrico Bambino Gesu ( Site 1301), Roma
- Russia (4):
  - Krasnoyarsk Regional Center for Prevention and Control of AIDS ( Site 1507), Krasnoyarsk, Krasnoyarsk Krai
  - Infectious Clinical Hospital #2 ( Site 1501), Moscow, Moscow
  - FGU Republican Clinical Infectious Hospital of Roszdrav ( Site 1500), Saint Petersburg, Sankt-Peterburg
  - Saratov Regional Clinical Center for Prophylaxis and Control of AIDS ( Site 1505), Saratov, Saratov Oblast
- South Africa (4):
  - Perinatal HIV Research Unit ( Site 1902), Johannesburg, Gauteng
  - Wits Reproductive Health and HIV Institute (WRHI) ( Site 1903), Johannesburg, Gauteng
  - Empilweni Services and Research Unit ( Site 1904), Johannesburg, Gauteng
  - King Edward Hospital ( Site 1900), Durban, KwaZulu-Natal
- Thailand (3):
  - Chulalongkorn University ( Site 1602), Bangkok, Bangkok
  - Siriraj Hospital ( Site 1601), Bangkok, Bangkok
  - Research Institute for Health Sciences ( Site 1603), Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pediatric participants who were ≥35 kg body weight and <18 years of age were recruited at 18 study sites located in Italy, Russian Federation, Thailand, South Africa, and the United States.
Groups:
- DOR/ISL: Virologically Suppressed Cohort: VS participants (had taken stable 2- or 3-drug combination ART for ≥3 months) pediatric participants with HIV-1 infection receive DOR/ISL for 96 weeks.
- DOR/ISL: Treatment Naive Cohort: TN participants with HIV-1 infection receive DOR/ISL for 96 weeks.
Period: Overall Study
Arm/Group | DOR/ISL: Virologically Suppressed Cohort | DOR/ISL: Treatment Naive Cohort
Started | 39 | 3
Completed | 22 | 2
Not Completed | 17 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Ongoing for safety monitoring | 14 | 1
Not completed — Excluded from results due to informed consent issue | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DOR/ISL: Virologically Suppressed Cohort | DOR/ISL: Treatment Naive Cohort | Total
Number analyzed (Participants) | 37 | 3 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.7 (2.2) | 15.7 (1.5) | 14.8 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 1 | 15
  Male | 23 | 2 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 35 | 3 | 38
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 3 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 0 | 20
  White | 8 | 0 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Drug Concentration-time Curve From 0 to 24 Hours Post-dose (AUC0-24) of Islatravir (ISL)
Description: The AUC0-24 of ISL in plasma was determined at steady state.
Time Frame: Pre-dose, and 0.5, 1, 2, 4, 8, 12, and 24 hours post-dose on Day 28
Population: A subset of VS participants was included in the Intensive PK Cohort, consisting of participants who complied with the protocol sufficiently to ensure data were likely to exhibit the effects of the study intervention on plasma PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*µmol/L
Arm/Group | DOR/ISL: Virologically Suppressed Cohort
Number analyzed (Participants) | 15
hr*µmol/L | 0.114 (28.6)

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of ISL
Description: The Cmax of ISL in plasma was determined at steady state.
Time Frame: Pre-dose, and 0.5, 1, 2, 4, 8, 12, and 24 hours post-dose on Day 28
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µmol/L
Arm/Group | DOR/ISL: Virologically Suppressed Cohort
Number analyzed (Participants) | 15
µmol/L | 0.0245 (53.4)

3. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of ISL
Description: The Tmax of ISL in plasma was determined at steady state.
Time Frame: Pre-dose, and 0.5, 1, 2, 4, 8, 12, and 24 hours post-dose on Day 28
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | DOR/ISL: Virologically Suppressed Cohort
Number analyzed (Participants) | 15
hours | 1.00 [0.50 to 4.00]

4. Primary Outcome: Apparent Plasma Terminal Half-life (t½) of ISL
Description: The t½ of ISL in plasma was determined at steady state.
Time Frame: Pre-dose, and 0.5, 1, 2, 4, 8, 12, and 24 hours post-dose on Day 28
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | DOR/ISL: Virologically Suppressed Cohort
Number analyzed (Participants) | 15
hours | 16.5 (70.0)

5. Primary Outcome: Apparent Total Clearance From Plasma (CL/F) of ISL
Description: The CL/F of ISL from plasma was determined at steady state.
Time Frame: Pre-dose, and 0.5, 1, 2, 4, 8, 12, and 24 hours post-dose on Day 28
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | DOR/ISL: Virologically Suppressed Cohort
Number analyzed (Participants) | 15
L/hr | 22.5 (28.6)

6. Primary Outcome: Apparent Volume of Distribution During Terminal Phase (Vz/F) of ISL
Description: The Vz/F of ISL was determined at steady state.
Time Frame: Pre-dose, and 0.5, 1, 2, 4, 8, 12, and 24 hours post-dose on Day 28
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | DOR/ISL: Virologically Suppressed Cohort
Number analyzed (Participants) | 15
Liters | 536 (61.1)

7. Primary Outcome: AUC0-last of ISL-triphosphate (ISL-TP) in Peripheral Blood Mononuclear Cells (PBMCs)
Description: The AUC0-24 of ISL-TP in PBMCs was determined at steady state.
Time Frame: Pre-dose, and 4 and 24 hours post-dose on Day 28
Population: A subset of VS participants was included in the Intensive PBMC PK Cohort, consisting of participants who complied with the protocol sufficiently to ensure data were likely to exhibit the effects of the study intervention on intracellular PBMC PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*pmol/10^6 cells
Arm/Group | DOR/ISL: Virologically Suppressed Cohort
Number analyzed (Participants) | 12
hr*pmol/10^6 cells | 52.3 (74.9)

8. Primary Outcome: Cmax of ISL-TP in PBMCs
Description: The Cmax of ISL-TP in PBMCs was determined at steady state.
Time Frame: Pre-dose, and 4, and 24 hours post-dose on Day 28
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/10^6 cells
Arm/Group | DOR/ISL: Virologically Suppressed Cohort
Number analyzed (Participants) | 12
pmol/10^6 cells | 2.87 (91.6)

9. Primary Outcome: C24 of ISL-TP in PBMCs
Description: The C24 of ISL-TP in PBMCs was determined at steady state.
Time Frame: 24 hours post-dose on Day 28
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/10^6 cells
Arm/Group | DOR/ISL: Virologically Suppressed Cohort
Number analyzed (Participants) | 12
pmol/10^6 cells | 2.05 (71.7)

10. Primary Outcome: Number of Participants Experiencing ≥1 Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to 24 weeks
Population: All participants who received ≥1 dose of study intervention are included.
Measure: Count of Participants; unit: Participants
Arm/Group | DOR/ISL: Virologically Suppressed Cohort | DOR/ISL: Treatment Naive Cohort
Number analyzed (Participants) | 37 | 3
Participants | 21 | 2

11. Primary Outcome: Number of Participants Discontinuing From Study Treatment Due to an AE
Description: as for outcome 10
Time Frame: Up to 24 weeks
Population: All participants who received ≥1 dose of study intervention are included.
Measure: Count of Participants; unit: Participants
Arm/Group | DOR/ISL: Virologically Suppressed Cohort | DOR/ISL: Treatment Naive Cohort
Number analyzed (Participants) | 37 | 3
Participants | 0 | 0

12. Secondary Outcome: Percentage of Virologically Suppressed (VS) Participants With HIV-1 Ribonucleic Acid (RNA) ≥50 Copies/mL
Description: The percentage of VS participants with HIV-1 RNA ≥50 copies/mL was determined at the central laboratory with an Abbott Real Time Polymerase Chain Reaction (PCR) assay with a lower limit of detection (LLOD) of 40 copies/mL.
Time Frame: Week 24
Population: Participants who were VS at baseline (on stable combination antiretroviral therapy [ART] for ≥3 months) and had data available are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DOR/ISL: Virologically Suppressed Cohort
Number analyzed (Participants) | 34
percentage of participants | 2.9 [0.1 to 15.3]

13. Secondary Outcome: Percentage of VS Participants With HIV-1 RNA <50 Copies/mL
Description: The percentage of VS participants with HIV-1 RNA <50 copies/mL will be determined at the central laboratory with an Abbott Real Time PCR assay with a LLOD of 40 copies/mL.
Time Frame: Week 24
Population: Participants who were VS at baseline (on stable combination ART for ≥3 months) and had data available are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DOR/ISL: Virologically Suppressed Cohort
Number analyzed (Participants) | 34
percentage of participants | 94.1 [80.3 to 99.3]

14. Secondary Outcome: Percentage of Treatment Naive (TN) Participants With HIV-1 RNA <50 Copies/mL
Description: The percentage of TN participants with HIV-1 RNA <50 copies/mL will be determined at the central laboratory with an Abbott Real Time PCR assay with a LLOD of 40 copies/mL.
Time Frame: Week 24
Population: Participants who were TN at baseline and had data available are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DOR/ISL: Treatment Naive Cohort
Number analyzed (Participants) | 1
percentage of participants | 100.0 [2.5 to 100.0]

15. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4+ (CD4+) T-cells in VS Participants
Description: CD4+ T-cell counts were measured by a central laboratory. Negative and positive results represent a decrease and increase, respectively, from baseline CD4+ T-cell counts.
Time Frame: Baseline (Day 1) and Week 24
Population: All VS participants who received ≥1 dose of study intervention and had data available are included.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | DOR/ISL: Virologically Suppressed Cohort
Number analyzed (Participants) | 33
cells/mm^3 | -112.1 [-175.8 to -48.4]

16. Secondary Outcome: Change From Baseline in CD4+ T-cells in TN Participants
Description: as for outcome 15
Time Frame: Baseline (Day 1) and Week 24
Population: TN participants who received ≥1 dose of study intervention and had baseline and Week 24 data available are included.
Measure: Number (95% Confidence Interval); unit: cells/mm^3
Arm/Group | DOR/ISL: Treatment Naive Cohort
Number analyzed (Participants) | 1
cells/mm^3 | 705.0 [NA to NA] — 95% CI not calculated due to n=1.

17. Secondary Outcome: Incidence of Viral Drug Resistance to DOR
Description: The number of participants with viral drug resistance to DOR was determined.
Time Frame: Up to 24 weeks
Population: Participants who received ≥1 dose of study intervention are included.
Measure: Count of Participants; unit: Participants
Arm/Group | DOR/ISL: Virologically Suppressed Cohort | DOR/ISL: Treatment Naive Cohort
Number analyzed (Participants) | 37 | 3
Participants | 0 | 0

18. Secondary Outcome: Incidence of Viral Drug Resistance to ISL
Description: The number of participants with viral drug resistance to ISL was determined.
Time Frame: Up to 24 weeks
Population: Participants who received ≥1 dose of study intervention are included.
Measure: Count of Participants; unit: Participants
Arm/Group | DOR/ISL: Virologically Suppressed Cohort | DOR/ISL: Treatment Naive Cohort
Number analyzed (Participants) | 37 | 3
Participants | 0 | 0

19. Secondary Outcome: Palatability of DOR/ISL Tablet
Description: The palatability of the DOR/ISL tablet (whole or split) was assessed with a modified 5-point facial hedonic scale. Responses ranged from 1 ("very bad") to 5 ("very good"). Data show the number of VS and TN participants responding at each score at the designated time points.
Time Frame: Baseline (Day 1), Week 4, and Week 24
Population: All VS and TN participants who received ≥1 dose of study intervention and have data available are included.
Measure: Count of Participants; unit: Participants
Arm/Group | DOR/ISL: Virologically Suppressed Cohort | DOR/ISL: Treatment Naive Cohort
Number analyzed (Participants) | 37 | 3
Participants
  Very Bad - Day 1 | 0 | 0
  Very Bad - Week 4 | 0 | 0
  Very Bad - Week 24: number analyzed (Participants) | 22 | 1
  Very Bad - Week 24 | 2 | 0
  Bad - Day 1 | 0 | 0
  Bad - Week 4 | 0 | 0
  Bad - Week 24: number analyzed (Participants) | 22 | 1
  Bad - Week 24 | 3 | 0
  Neither good or bad - Day 1 | 12 | 0
  Neither good or bad - Week 4 | 11 | 0
  Neither good or bad - Week 24: number analyzed (Participants) | 22 | 1
  Neither good or bad - Week 24 | 8 | 0
  Good - Day 1 | 9 | 2
  Good - Week 4 | 11 | 2
  Good - Week 24: number analyzed (Participants) | 22 | 1
  Good - Week 24 | 5 | 1
  Very Good - Day 1 | 16 | 1
  Very Good - Week 4 | 15 | 1
  Very Good - Week 24: number analyzed (Participants) | 22 | 1
  Very Good - Week 24 | 4 | 0

20. Secondary Outcome: Acceptability of DOR/ISL Tablet
Description: The acceptability of the DOR/ISL tablet (whole or split) was assessed. Acceptability was assessed by monitoring for refusing the tablet, throwing up or spitting out the tablet, and gagging on the tablet. Data show the number of VS and TN participants responding at each score at the designated time points.
Time Frame: Baseline (Day 1), Week 4, and Week 24
Population: All VS and TN participants who received ≥1 dose of study intervention and have data available are included.
Measure: Count of Participants; unit: Participants
Arm/Group | DOR/ISL: Virologically Suppressed Cohort | DOR/ISL: Treatment Naive Cohort
Number analyzed (Participants) | 37 | 3
Participants
  Refusing - Day 1 | 0 | 0
  Refusing - Week 4 | 0 | 0
  Refusing - Week 24: number analyzed (Participants) | 22 | 1
  Refusing - Week 24 | 0 | 0
  Throwing Up/Spitting Out - Day 1 | 0 | 0
  Throwing Up/Spitting Out - Week 4 | 0 | 0
  Throwing Up/Spitting Out - Week 24: number analyzed (Participants) | 22 | 1
  Throwing Up/Spitting Out - Week 24 | 0 | 0
  Gagging - Day 1 | 0 | 0
  Gagging - Week 4 | 0 | 0
  Gagging - Week 24: number analyzed (Participants) | 22 | 1
  Gagging - Week 24 | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 16 months
Description: All-cause mortality was assessed in all randomized participants. Adverse events (AEs) and serious AEs (SAEs) were assessed in all treated participants.
Groups:
- DOR/ISL: Virologically Suppressed Cohort Extended Monitoring: VS participants with confirmed protocol-specified decreases in CD4+ T-cell and/or total lymphocyte counts are in extended safety monitoring after switching to non-study ART.
- DOR/ISL: Treatment Naive Cohort Extended Monitoring: TN participants with confirmed protocol-specified decreases in CD4+ T-cell and/or total lymphocyte counts are in extended safety monitoring after switching to non-study ART.
Arm/Group | DOR/ISL: Virologically Suppressed Cohort | DOR/ISL: Treatment Naive Cohort | DOR/ISL: Virologically Suppressed Cohort Extended Monitoring | DOR/ISL: Treatment Naive Cohort Extended Monitoring
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/3 | 0/14 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/37 | 0/3 | 0/14 | 0/1
Other Adverse Events (participants affected / at risk) | 13/37 | 2/3 | 12/14 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DOR/ISL: Virologically Suppressed Cohort (N=37) | DOR/ISL: Treatment Naive Cohort (N=3) | DOR/ISL: Virologically Suppressed Cohort Extended Monitoring (N=14) | DOR/ISL: Treatment Naive Cohort Extended Monitoring (N=1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DOR/ISL: Virologically Suppressed Cohort (N=37) | DOR/ISL: Treatment Naive Cohort (N=3) | DOR/ISL: Virologically Suppressed Cohort Extended Monitoring (N=14) | DOR/ISL: Treatment Naive Cohort Extended Monitoring (N=1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Vaccination site pain (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 3 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 4 (7) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 2 (4) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 3 (4) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (4) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post-acute COVID-19 syndrome (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT04295772/Prot_SAP_000.pdf